CLINICAL TRIAL: NCT03033472
Title: Effect of Preoperative Single-dose Clindamycin on Postoperative Endodontic Pain in Patients With Symptomatic Apical Periodontitis: A Randomized Controlled Trial
Brief Title: Effect of Preoperative Clindamycin on Postoperative Endodontic Pain
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nermeen Saeed Abdel Ghany El Sedawy, principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEBC-CU-2017-01-09
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Symptomatic Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind (Subject, Caregiver, Investigator, Outcomes Assessor) Primary Purpose: Treatment

ARMS (2):
- Clindamycin (Experimental): 600 mg of Clindamycin orally 30 minutes before root canal treatment
  Interventions: Drug: 600 mg Clindamycin orally
- Placebo (Placebo Comparator): placebo 30 minutes Orally before treatment
  Interventions: Drug: Oral Placebo

INTERVENTIONS:
Drug: 600 mg Clindamycin orally — 600 mg Clindamycin orally 30 minutes before treatment
  Arms: Clindamycin
Drug: Oral Placebo — Oral Placebo 30 minutes before treatment
  Arms: Placebo

SUMMARY:
The aim of this prospective, randomized, placebo controlled study is to evaluate the effect of clindamycin on post-operative pain and swelling in adult patient with symptomatic apical periodontitis.

DETAILED DESCRIPTION:
Medical and dental history will be obtained from all patients participating in this trial. Clinical and radiographic evaluation for each tooth included in this study will be recorded.

Clinical diagnosis of symptomatic apical periodontitis is to be confirmed.

Before root canal treatment, eligible participants will be randomly assigned to one of the following groups: experimental group (taking 600 mg of clindamycin orally) or control group (taking placebo ) 30 minutes before the start of the treatment. Single-visit root canal treatment will be performed.

Each patient will receive a 7-day diary to record postoperative pain and swelling.In case of pain, the participant will be instructed to take an analgesic. Post-operative pain will be measured as a primary outcome on 11-point scale (NRS) at the following time points: 6, 12, 24, 48, 72 hours and 7 days. The occurrence of swelling will be reported by participant as a secondary outcome

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic apical periodontitis and do not have evidence of spreading infection or systemic involvement.
2. Mandibular posterior teeth.
3. Patients in good health.
4. Patients who can understand pain scales (NRS).
5. Patients able to sign informed consent.

Exclusion Criteria:

1. Patients who have draining sinus tract.
2. Retreatment cases
3. Patients with weeping canals.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | Up to 7 days after endodontic treatment
  Post-operative pain will be measured by a numerical rating scale (NRS)

SECONDARY OUTCOMES:
Swelling | 7 days
  The occurrence of Swelling will be measured by a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nermeen SA El Sedawy, Post Graduate, Principal Investigator — Cairo University; Suzan AW Wanees, PhD, Study Chair — Cairo Univertsity; Shaimaa Gawdat, PhD, Study Director — Cairo University

REFERENCES:
- [Result] Cope A, Francis N, Wood F, Mann MK, Chestnutt IG. Systemic antibiotics for symptomatic apical periodontitis and acute apical abscess in adults. Cochrane Database Syst Rev. 2014 Jun 26;(6):CD010136. doi: 10.1002/14651858.CD010136.pub2. PMID 24967571
- [Result] Lindeboom JA, Frenken JW, Valkenburg P, van den Akker HP. The role of preoperative prophylactic antibiotic administration in periapical endodontic surgery: a randomized, prospective double-blind placebo-controlled study. Int Endod J. 2005 Dec;38(12):877-81. doi: 10.1111/j.1365-2591.2005.01030.x. PMID 16343114